CLINICAL TRIAL: NCT01959087
Title: Single Port Colic Laparoscopic Surgery - THE TRUE TRIAL
Brief Title: Single Port Colic Laparoscopic Surgery
Acronym: TRUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P111112
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Colonic Neoplasms; Crohn's Disease; Diverticulitis
Keywords: Single port surgery; Colonic surgery; Postoperative morbidity; Postoperative outcomes
MeSH Terms: conditions — Colonic Neoplasms; Crohn Disease; Diverticulitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Single port surgery (Experimental): Surgery with single port
  Interventions: Procedure: single port surgery; Procedure: Multiport surgery
- 2: Multiport surgery (Active Comparator): Surgery with multiport
  Interventions: Procedure: Multiport surgery

INTERVENTIONS:
Procedure: single port surgery — Single port surgery can be converted in multiport surgery if necessary
  Arms: 1: Single port surgery
Procedure: Multiport surgery

SUMMARY:
This study aims to compare the results of colonic surgery performed by single and multiport laparoscopy.

DETAILED DESCRIPTION:
The aim of this study is to compare surgical results of colonic resection performed by single port and multiport laparoscopic approaches. Primary endpoint is the length of postoperative hospital stay. Secondary endpoints include postoperative mortality, postoperative morbidity, conversion rates, postoperative recovery, aesthetic results, postoperative pain, and costs

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Colonic resection performed for benign or malignant colonic neoplasm, Crohn's disease, or diverticulitis
* Informed consent signed
* Social Insurance

Exclusion Criteria:

* Digestive stoma in place or planned during the intervention
* Body mass index > 30 kg/m2
* History of previous laparotomy, except Mc Burney, Pfannenstiel ou subcostal
* Subtotal colectomy
* Transverse colectomy
* Proctectomy or total coloproctectomy
* Synchronous metastasis
* Preoperative suspicion of T4 colorectal cancer
* Emergency procedure
* Associated resection (except appendectomy or liver biopsy)
* Pregnancy or current breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Length of postoperative hospital stay | 30 days
  Theoretical duration of hospitalization (from the day of the surgery to the theoretical date of discharge

SECONDARY OUTCOMES:
Operative mortality | 30 days
  Operative mortality rate; Overall morbidity rate at 30 days postoperatively including infectious and noninfectious morbidity according to the DINDO classification; Rates of incisional herniation, occlusion, rehospitalization related to the surgical procedure and reintervention until J180; Actual hospital stay;
Post-operative morbidity | Day 30
Conversion rates | Day 1
Pathologic results | Day 180
Postoperative recovery | 30 days
Postoperative pain | 6 days
Aesthetic results | 180 days
Costs | Day 180
Lenght of true hospitalization stay | 30 days
Technical feasability | Day 1
Post-operative quality of life | Day 180
  SF-36 and GIQLI

CONTACTS AND LOCATIONS:
Overall Officials: Yves PANIS, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Chirurgie Colorectale, Clichy, Île-de-France Region, France

REFERENCES:
- [Derived] Maggiori L, Tuech JJ, Cotte E, Lelong B, Denost Q, Karoui M, Vicaut E, Panis Y. Single-incision Laparoscopy Versus Multiport Laparoscopy for Colonic Surgery: A Multicenter, Double-blinded, Randomized Controlled Trial. Ann Surg. 2018 Nov;268(5):740-746. doi: 10.1097/SLA.0000000000002836. PMID 30303873